CLINICAL TRIAL: NCT02482922
Title: Feasibility of an Interval Exercise and Nutrition Intervention to Reduce Cardiovascular Disease Risk
Brief Title: Feasibility of an Interval Exercise and Nutrition Intervention to Reduce Cardiovascular Disease Risk Factors
Acronym: IETnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Abbie Smith-Ryan, PhD, Assistant Professor, University of North Carolina, Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13-3515
Record Dates: First submitted 2015-06-22; First posted 2015-06-26 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Pre-Diabetic; Overweight; Obesity
Keywords: feasibility studies; intervention; Pre-Hypertensive; Pre-Hyperlipidemia
MeSH Terms: conditions — Glucose Intolerance; Overweight; Obesity | interventions — Exercise; Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IET and Nutrition (Experimental): 3 times per week of interval exercise training Once daily meal replacement
  Interventions: Other: Exercise & Dietary Supplement

INTERVENTIONS:
Other: Exercise & Dietary Supplement

SUMMARY:
Purpose : Test the feasibility (acceptability, adherence) of a home-based interval exercise training (IET) and nutrition program, as well as its preliminary effects on resting heart rate, blood pressure, fasting glucose, HDL, cholesterol, weight and percent body fat, among primary care patients who have at least one risk factor for cardiovascular disease (CVD).

Participants : 30 patients who receive care from the University of North Carolina (UNC) Family Medicine Center (FMC) and meet the inclusion criteria defined below (i.e. general FMC patients, not diagnosed with severe illness), will be enrolled to test the feasibility of the home-based interval exercise and nutrition program.

Procedures (methods): A home-based IET and nutrition program will be piloted in 2 phases. In Phase I, 15 patients will be enrolled into the program, which will take approximately 3 months. At baseline, data will be collected on age, height, weight, resting heart rate, blood pressure, fasting glucose, hemoglobin A1c, fasting lipids, cholesterol, insulin, percent body fat, cardiovascular fitness, and use a series of questionnaires to evaluate mood, sleep, hunger, and quality of life. At closeout, the investigators will measure patients' adherence to each component of the intervention. In Phase II, an additional 15 new patients will be enrolled in either the identical protocol, or a slightly modified intervention (if necessary based upon our results from Phase I). All patients will have the same variables measured at baseline during their study visit at 3, 6 and 12 months after enrollment into the study.

ELIGIBILITY:
Inclusion Criteria:

Patients are:

1. > 18-85 years;
2. receive primary care in the FMC (> 1 visit during the previous year); and
3. have ≥1 risk factor or developing risk factors for CVD (blood pressure >130/85 mmHG, BMI >25 kg/m2(or ~20 lbs overweight), Fasting glucose >110 mg/dl, OR 4) HDL <30) (all identified via medical record)

Exclusion Criteria:

1. those for whom exercise and/or diet are contraindicated (e.g., scheduled for arthroplasty) or who are at risk of death in the next year (e.g., Class IV heart failure, end-stage renal disease).
2. those taking medication for diabetes, blood pressure, and lipids for more than 2 years.
3. pregnant or planning on becoming pregnant within the next year.
4. Allergic to any ingredient in the nutritional meal replacement.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-05; Primary Completion 2016-05 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Number of participants that complete exercise program | 3 months
Number of participants that complete nutrition program | 3 months
Number of exercise sessions completed | 3 months
Number of days nutrition program followed | 3 months

SECONDARY OUTCOMES:
Change in Cardiorespiratory Fitness at 3 months, 6 months, and 12 months | 3 months, 6 months, 12 months
Change in fat mass at 3 months, 6 months, and 12 months | 3 months, 6 months, 12 months
Change in lean mass at 3 months, 6 months, and 12 months | 3 months, 6 months, 12 months
Change in blood lipids at 3 months, 6 months, 12 months | 3 months, 6 months, 12 months
Change in hemoglobin A1c at 3 months, 6 months, 12 months | 3 months, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Abbie Smith-Ryan, PhD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina Family Medicine Center, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Smith-Ryan AE, Weaver MA, Viera AJ, Weinberger M, Blue MNM, Hirsch KR. Promoting Exercise and Healthy Diet Among Primary Care Patients: Feasibility, Preliminary Outcomes, and Lessons Learned From a Pilot Trial With High Intensity Interval Exercise. Front Sports Act Living. 2021 Jul 16;3:690243. doi: 10.3389/fspor.2021.690243. eCollection 2021. PMID 34337406